CLINICAL TRIAL: NCT01981928
Title: A Phase 1, Randomized, Subject- and Investigator-blinded, Sponsor-unblinded, Placebo-controlled, Parallel Group Study to Assess the Safety, Tolerability and Pharmacokinetics of Single Ascending Oral Doses of ASP7962, Including a Food-effect Evaluation in Healthy Subjects
Brief Title: A Clinical Trial to Investigate Safety and Tolerability of ASP7962 in Healthy Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 7962-CL-0001; 2013-001738-16 (EudraCT Number)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Safety; Tolerability; Pharmacokinetics of ASP7962
Keywords: Phase 1; Healthy Subjects; Safety; Tolerability; Pharmacokinetics; Single Ascending Oral Dose; Food Effect

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP7962 (Experimental): Each dose level group will include 8 subjects, of which 6 will be randomized to receive active ASP7962
  Interventions: Drug: ASP7962
- Placebo (Placebo Comparator): Each dose level group will include 8 subjects, of which 2 will be randomized to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP7962 — Oral
  Arms: ASP7962
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The purpose of the study is to see how safe the study drug is and how well it is tolerated after dosing. The study will also investigate how the study drug is taken up, metabolized (chemically broken down), distributed through the body and excreted. A further aim is to look at how this process is possibly altered by food by giving the study drug in the presence and absence of meals.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body mass index (BMI) range of 18.5 - 30.0 kg/m2, inclusive. The subject weighs at least 50 kg. [screening]
* Female subject must be of non-childbearing potential:postmenopausal (defined as at least 1 year without any menses) prior to screening, or documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening).
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continue throughout the clinical study period and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the clinical study period and for 90 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while in this clinical study.

Exclusion Criteria:

* Subject has a known or suspected hypersensitivity to ASP7962 or any components of the formulation used.Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy, as judged by the Medical Investigator.
* Subject has any clinically significant abnormality following the Investigator's review of the physical examination, ECG and clinical study protocol-defined clinical laboratory tests at screening or on admission to the clinical unit on day -1.
* Subject regularly uses any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the clinical unit on day -1.
* Subject had any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to admission to the clinical unit on day -1.
* Subject participated in any interventional clinical study or has been treated with any investigational drugs within 90 days or 5 half-lives whichever is longer, prior to the initiation of screening
* Subject has a history of suicide attempt or suicidal behavior. Any recent suicidal ideation within the last 3 months (a level of 4 or 5 for any 1 item on the scale), or who are at significant risk to commit suicide, as judged by the Investigator using the C-SSRS at screening and on admission to the clinical unit on day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety assessed by: clinical laboratory tests, vital signs, Electrocardiogram (ECG), Adverse Events (AEs), real time and continuous cardiac monitoring, orthostatic challenge test, and C-SSRS | Day -1 through End of Study Visit (7 to 14 days after (early) discharge from the clinical unit (only after the second treatment period for subjects required to return for the food-effect part of the clinical study))
  Day 1 to End of Study Visit: Routine clinical laboratory tests (hematology, biochemistry [additionally including testosterone, luteinizing hormone {LH}, follicle-stimulating hormone {FSH}, inhibin b, sex hormone-binding globulin {SHBG}] and urinalysis), Vital Signs, ECG, A Es Day 1: Real-time cardiac monitoring Day 1 to Day 2: Continuous cardiac monitoring and orthostatic challenge test Day -1 and End of Study Visit: C-SSRS for suicidality risk

SECONDARY OUTCOMES:
Pharmacokinetics of ASP7962 in plasma and urine | Day 1 to Day 7
  Measurement of ASP7962 in plasma and urine under fasted and fed conditions. Plasma: AUCinf, AUCinf,u, AUClast, AUClast,u, Cmax, Cmax,u, CL/F, CLu/F, fu, tlag, tmax, t½, Vz/F, Vz,u/F Urine: Aelast, Aeinf, Aelast%, Aeinf%, CLR, CLR,u

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Parexel Early Phase Clinical Unit London, London, United Kingdom